CLINICAL TRIAL: NCT04694261
Title: Resilience, Depression And Anxiety Among Pregnant Women In Pakistan: Development And Testing Of Intervention
Brief Title: Development and Evaluation of SM-ART Intervention (SM-ART)
Acronym: SM-ART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: University Ghent (Other)
Responsible Party: Principal Investigator, Shireen Shehzad Bhamani, Assistant Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5312-SON-ERC-18.; 70345 (182015SONAM) (Other Grant/Funding Number: University Research Council)
Record Dates: First submitted 2020-12-31; First posted 2021-01-05 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Perinatal Depression; Resilience; Anxiety; Marital Conflict
Keywords: Resilience; Perinatal mental health; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: The assessments will be carried out parallel in the intervention and the control arm.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessors will not be aware about the allocation of assignments between intervention and control arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SM-ART Intervention (Experimental): Intervention group will receive SM-ART module training along with the flyers on resilience building tips.
  Interventions: Behavioral: SM-ART
- Control Group (No Intervention): Control group will only receive flyer on resilience building tips

INTERVENTIONS:
Behavioral: SM-ART — Intervention is a group based training delivered by midwives on SM-ART module. These training will consist of 6 sessions, one per week for 90 to 120 minutes each.
  Arms: SM-ART Intervention

SUMMARY:
The approach of this intended research is to help pregnant women practice constructive coping and proactive skills that focus on positive adaptation for safe motherhood through our developed intervention.

The objective of this two phases Randomized Control Trial is to develop contextually based "SM-ART" intervention [Safe Motherhood ART: Accessible Resilience Training] and evaluate the effectiveness of "SM-ART" intervention in a sample of pregnant women living in low socioeconomic urban areas of Karachi, Pakistan.

It is hypothesized that the SM-ART intervention will enhance resilience and marital harmony and decrease symptoms of depression, anxiety in pregnant women.

DETAILED DESCRIPTION:
The prevalence of perinatal depression and anxiety in South Asia are among the highest in the world. In Pakistan, approximately 18% to 60% of women experienced depressive symptoms at some point during their pregnancy. Early intervention for the management of mental illness in pregnancy is imperative as the effects of perinatal mental ill-health is not only limited to mothers but also can negatively impact child health outcomes. In a public health context, positive psychological interventions should be promoted as it reduces the burden of treatment, and enhance cost effective approaches in resource poor countries such as Pakistan.

As in Pakistan, no program has been planned and tested to enhance the positive psychological wellbeing among pregnant women that is based on individual strengths, that can be learnt, sustained and low cost as well. Hence, this study aims to facilitate pregnant women in practicing constructive coping and proactive skills which will help them to focus more on the positive approach of life rather than looking for the negative situations that is carried out in their daily lives.

The study will carried out in two phases:

Phase I: The objective of phase one is study is to develop "SM-ART" intervention [Safe Motherhood ART: Accessible Resilience Training]

Phase II: The objective of phase two is to test the effectiveness of "SM-ART" intervention [Safe Motherhood ART: Accessible Resilience Training] to improve resilience, marital harmony and decrease depression and pregnancy related anxiety in a sample of pregnant women presenting to Koohi Goth Hospital of Karachi, Pakistan

ELIGIBILITY:
Inclusion Criteria:

1. All participants should provide written consent, be 18+ years of age
2. All participants should be currently married at a gestational age of 12 to 30 weeks: by 12th week, pregnancy is confirmed, they do visit health clinic and upper bar is set to 30 weeks so there should be adequate time to provide the intervention and observe the effectiveness.
3. Participants should speak and understand urdu, as all our assessments and intervention will be in local language.

Exclusion Criteria:

Participants with a history of mental illness and/or physical illness will be excluded as will those taking antianxiety, antidepressant, anti psychotic medication.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 200 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Resilience Score | Baseline ( at the time of enrolment) and Post assessment (within two weeks of intervention)
  Resilience Scale 14: This is a 14 items scale which score ranges from 14 to 98. It represent all five characteristics of resilience: A purposeful life, Perseverance, Equanimity, Self-reliance and Existential aloneness. A higher total score indicates higher resilience. The scale also have cutoffs as well. The scale is validated in Pakistani population by the current study principle investigator.

SECONDARY OUTCOMES:
Change in Depression score | Baseline ( at the time of enrolment) and Post assessment (within two weeks of intervention)
  Edinburgh Postnatal Depression Scale (EPDS):10-item; range 0-30, cut-off 13; across 15 countries including some LMIC Cronbach's α=.73-.87; 3 to 12 week test-retest=.53-.74) measures depression.
Change in Pregnancy related Anxiety score | Baseline ( at the time of enrolment) and Post assessment (within two weeks of intervention)
  Pregnancy-related anxiety scale-revised, (10 items; range 10-40; Cronbach's α=.78) evaluates feelings about health during pregnancy, health of fetus/infant, and labour and delivery.
Change in Marital Adjustment score | Baseline ( at the time of enrolment) and Post assessment (within two weeks of intervention)
  Locke Wallace Marital Adjustment Test (15 Items) It focuses on the aspects like participation in shared activities, display of affection and spouse agreement on important matters related to marital adjustment. It is an extensively used self-report measure of adjustment in marriage. The scale scores range from 2-158. A score less than 100 indicate marital distress.

CONTACTS AND LOCATIONS:
Overall Officials: Shireen S Bhamani, PhD Student, Principal Investigator — Aga Khan University School of Nursing & Midwifery; Olivier Degomme, Study Chair — University Ghent; An-Sofie Van Parys, Study Director — University Ghent; David Arthur, Study Director — Aga Khan University
Locations (1):
- Koohi Goth Women Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data will be analyzed using unique identifier and only the password protected data may be shared with the supervisory team of researchers.

REFERENCES:
- [Derived] Bhamani SS, Van Parys AS, Arthur D, Letourneau N, Wagnild G, Degomme O. Promoting mental wellbeing in pregnant women living in Pakistan with the Safe Motherhood-Accessible Resilience Training (SM-ART) intervention: a randomized controlled trial. BMC Pregnancy Childbirth. 2024 Jun 29;24(1):452. doi: 10.1186/s12884-024-06629-2. PMID 38951777